CLINICAL TRIAL: NCT00071682
Title: Early Identification of Adverse Reactions to Herbs
Brief Title: Evaulation of Interaction Between Herbal Products and Anticoagulants
Status: Withdrawn | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: K08AT001338-01 (NIH); K08AT001338-01 (NIH)
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Coagulation Disorders
Keywords: herbal medicine; alternative medicines; anticoagulation; side effects; bleeding; clotting
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage; Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the use of herbal products interferes with normal anticoagulation, leading to either excessive thinning of the blood and bleeding problems or inadequate thinning of the blood and clotting problems. Many patients who are on long term anticoagulation, or blood thinning, for a variety of medical problems, also take herbal products. It is not yet known whether use of herbal products interferes with this anticoagulation, and puts patients at risk for bleeding or clotting. This study will carefully monitor patients who are taking herbs and anticoagulants to determine if their laboratory tests show signs of being affected by the herbs. The study will ask all patients about their herbal product use, so all reported herbs will be included and monitored.

ELIGIBILITY:
Inclusion criteria:

* Taking longer-term (>6 months) anticoagulation
* Enrolled in one of Kaiser Permanente Northern California anticoagulation clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bent, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States